CLINICAL TRIAL: NCT07060404
Title: Pharmacokinetics of Primaquine and Tafenoquine in Lactating Women - Towards Equitable Radical Cure of Vivax Malaria
Brief Title: Postpartum 8-aminoquinoline Breast Milk Study
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Curtin University (Other)
Collaborators: Menzies School of Health Research (Other); Papua New Guinea Institute of Medical Research (Other Government)
Responsible Party: Principal Investigator, Brioni Moore, Associate Professor, Curtin University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: RES68007
Record Dates: First submitted 2025-06-11; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Drug Pharmacokinetics in Healthy Volunteers
Keywords: primaquine; tafenoquine; vivax malaria; pharmacokinetics; postpartum; lactation; infant exposure
MeSH Terms: conditions — Malaria, Vivax; Breast Feeding | interventions — Food; Water; Primaquine; tafenoquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group1 - control (No Intervention): Participants will receive no intervention at time of delivery. As per standard care in PNG, each participant will receive primaquine at 6-months postpartum (completion of study procedures).
- Group 2 - PQ14 (Experimental): Daily oral primaquine as 0.5 mg/kg per day for 14 days, taken with food and water
  Interventions: Drug: Daily primaquine (0.5 mg/kg per day) for 14 days given with food food and water
- Group 3 - PQ7 (Experimental): Daily oral primaquine 1 mg/kg per day for 7 days, taken with food and water
  Interventions: Drug: Daily primaquine 1 mg/kg per day for 7 days given with food and water
- Group 4 - TQ (Experimental): Single dose tafenoquine as 300mg taken with food and water
  Interventions: Drug: Single-dose tafenoquine given with food and water to prevent gastrointestinal discomfort

INTERVENTIONS:
Drug: Daily primaquine (0.5 mg/kg per day) for 14 days given with food food and water — Women will receive daily doses of PQ (0.5 mg/kg per day) for 14 days at a total treatment dose of 7 mg/kg PQ. All doses will be to the nearest full tablet, with food and water to prevent gastrointestinal discomfort, as directly observed treatment. Women vomiting within 30 minutes of administration of any dose will be re-treated.
  Other Names: Primacin; Primaquine phosphate
  Arms: Group 2 - PQ14
Drug: Daily primaquine 1 mg/kg per day for 7 days given with food and water — Women will receive daily doses of PQ (1 mg/kg per day) for 7 days at a total treatment dose of 7 mg/kg PQ. All doses will be to the nearest full tablet, with food and water to prevent gastrointestinal discomfort, as directly observed treatment. Women vomiting within 30 minutes of administration of any dose will be re-treated.
  Other Names: Primacin; Primaquine phosphate
  Arms: Group 3 - PQ7
Drug: Single-dose tafenoquine given with food and water to prevent gastrointestinal discomfort — Women will receive a single dose of 300mg tafenoquine. Treatment will be given with food and water to prevent gastrointestinal discomfort, as directly observed treatment. Women vomiting within 30 minutes of administration of any dose will be re-treated.
  Other Names: Tafenoquine succinate; Kodatef
  Arms: Group 4 - TQ

SUMMARY:
In Papua New Guinea, administration of primaquine (PQ) or tafenoquine (TQ) to breastfeeding mothers is contraindicated during the first six months postpartum, when infants are recommended to be exclusively breastfed, because of a lack of comprehensive pharmacokinetic data on PQ/TQ neonatal and infant exposure via breast milk. The therapeutic restriction of PQ/TQ use in lactating women during the first six months postpartum effectively translates into ~10% of females being excluded from radical cure in endemic areas at any time. This is because many at risk women live in remote areas, are frequently lost to follow-up, or may have conceived again before they reattend. As a result, radical cure is rarely achieved and women are exposed to recurrent infections and cumulative risk of anaemia. Relapses may occur for years, placing subsequent pregnancies at risk and perpetuating intergenerational failure of fetal growth. They also contribute to malaria transmission, thus household and community exposure to vivax malaria.

The goal of the present study is to determine how much PQ/TQ is transferred to a suckling baby, if a mother receives a treatment course of PQ/TQ at time of delivery. We also want to confirm that this treatment is safe and has no major side effects for babies in Papua New Guinea.

The study Interventions areas follows: Group 1 - Participants receive PNG standard of care; PQ given 6-months postpartum; Group 2 - Participants receive a 14-day treatment regimen of PQ, at the standard dose prescribed in PNG for vivax radical cure (0.5 mg/kg/day for 14 days); Group 3 - Participants receive an accelerated high-dose 7-day treatment regimen of PQ, as per current WHO recommendations (1.0 mg/kg/day for 7 days); Group 4 - Participants receive a single dose of 300mg tafenoquine.

All participants will be monitored for a total duration of 6 months, with the safety, tolerability, pharmacokinetics and preliminary relapse efficacy of PQ/TQ evaluated at standardised time points over this period (Day 0, 1, 3, 6, 8, 15, 20, 28, and Month 2, 3, 4, 5 and 6). At each of these time points, participants will be asked to describe any symptoms they may be experiencing, participate in a medical examination, and provide a blood and breast milk sample for drug analysis and safety (biochemistry and haematology testing). The investigators will also collect a small blood sample (heel prick) from the infant to measure drug concentrations and safety testing.

DETAILED DESCRIPTION:
Global malaria eradication requires universal and equitable access to effective antimalarial treatment. More than 2.5 billion people are at risk of infection with Plasmodium vivax. Unlike falciparum malaria, P. vivax forms dormant liver-stage parasites (hypnozoites) that can reactivate (relapse) causing recurrent febrile illness after the initial infection. Women are at increased risk of vivax malaria during pregnancy and postpartum, when they are at higher risk of P. vivax infections than P. falciparum malaria. Over 80% of these infections are relapses, rather than new infections but pregnant and lactating women cannot be treated with the available anti-relapse drugs. This is because the 8-aminoquinolones, primaquine (PQ) and tafenoquine (TQ), can cause potentially life-threatening haemolysis in glucose-6-phosphate dehydrogenase (G6PD)-deficient babies, and there is concern that the drugs are transferred in breast milk. If anti-relapse treatment could be given immediately on delivery and before discharge, it would dramatically reduce the risk of vivax relapses which currently affect ~10% of women in countries like Papua New Guinea (PNG).

This study aims to accelerate maternal access to PQ/TQ by confirming minimal transfer of PQ or TQ not only in mature breast milk (>2 weeks postpartum; current data available from a pharmacokinetic (PK) study in Thailand), but also in colostrum and transitional breast milk in the first two weeks after birth. Generating PK data for TQ is also critical. Maternal treatment could then be initiated before hospital discharge to prevent postpartum relapses and maximise benefit for health outcomes and malaria control.

This open-label study has the following objectives and hypothesis:

Primary Objective: To determine the transfer of primaquine (and primary metabolite carboxyprimaquine) and tafenoquine in breast milk (colostrum and transitional milk) and determine associated relative infant exposure.

Secondary objectives include; i) To compare haematological and hepatorenal indices in exposed and unexposed mother-infant pairs as a measure of safety, and ii) to assess maternal tolerability of early postpartum primaquine (PQ) and tafenoquine (TQ) treatment.

Hypothesis: i) Negligible concentrations of PQ and TQ will be detected in colostrum and transitional milk, or breastfed infants, when mothers are treated with PQ or TQ and ii) Maternal administration of therapeutic doses of PQ or TQ immediately after birth does not result in clinically significant haematological or hepatorenal changes in breastfed neonates.

To do this, once eligibility is confirmed, and appropriate informed consent obtained, a sample of 60 postpartum mother-infant pairs will be recruited into one of four study treatment groups (n=15 per treatment group).

Due to the nature of the research, a conservative approach will be taken to treatment allocation, with groups (n=15) of participants to be allocated treatment doses in a stepwise design as follows: Group 1 - non-intervention (control) group; Group 2 - PQ14 (0.5 mg/kg/day for 14 days); Group 3 - PQ7 (1 mg/kg/day for 7 days); and Group 4 - TQ (300 mg single dose).

Review of mother and neonate for safety and PK procedures across all groups will be scheduled on days 0, 1, 3, 6, 8, 15, 20 and 28 (and 56 for Group 4). At each scheduled time point a symptom questionnaire (capturing both maternal symptoms and the mother's observations of her child) will be conducted, along with a physical examination of both mother and infant. Samples for PK (maternal venous blood, maternal dried blood spot, fore- and hind-breast milk, infant dried blood spot) and safety assessment (haemoglobin, methaemoglobin, hepatorenal biochemistry) will also be collected at specified time points to confirm safety and characterise the transfer and PK profile of PQ/TQ in breast milk and associated infant exposure.

After completion of procedures (Day 28 for Groups 1-3 and Day 59 for Group 4) standardized review of each mother and infant will be conducted monthly for 6 months after initial treatment to monitor P. vivax recurrence and other indicators of maternal and infant health. These study review visits will be timed to coincide with the national infant immunisation schedule at 1, 2, 3 and 6 months. Examination of the infant by study staff will complement assessment of developmental milestones, and maternal assessment could include family planning.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Both mother and infant have G6PD activity >70% (normal activity; SD Biosensor)
3. They have no significant co-morbidity
4. Delivered a live singleton baby within past 48-hours
5. Rapid diagnostic test negative for malaria
6. No history of hypersensitivity to 8-aminoquinoline drugs
7. Plan to exclusively breastfeed for at least two months
8. History of vivax malaria (as per health book)
9. They can attend follow-up assessments for the duration of the study

Exclusion Criteria:

1. Either mother/infant have G6PD activity <70% (SD Biosensor)
2. Either mother/infant have significant co-morbidity
3. Mother did not deliver a live singleton within past 48-hours
4. Mother/infant are rapid diagnostic test positive for malaria
5. Mother has a history of hypersensitivity to 8-aminoquinoline drugs
6. Mother does not plan to exclusively breastfeed for at least two months
7. Mother does not have a history of vivax malaria (as per health book)
8. Cannot or are not willing to attend follow-up assessments for the duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females as required to be lactating postpartum women
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic: Distribution half -life | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ)
  Pharmacokinetic parameters of primaquine (PQ) (and primary metabolite carboxyprimaquine) and tafenoquine (TQ) in breast milk (colostrom and transitional milk) to determine relative infant exposure. Based on drug concentrations determined from venous blood samples (mothers) and heel prick samples (infants) collected at baseline (Day 0) 1, 3, 6, 8,15, 20 and 28 (and 56 for Group 4).
Pharmacokinetic: Termination elimination half-life | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ).
Pharmacokinetic: Absorption half-life | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ).
Pharmacokinetics: Clearance | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ).
Pharmacokinetics: Volume of distribution | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ).
Pharmacokinetics: Maximal concentration | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ).
Pharmacokinetics: Area under concentration-time curve | Group 2 and 3: 28 days after first drug dose (PQ) and Group 4: 56 days after drug administration (TQ).

SECONDARY OUTCOMES:
Safety: Change in haemoglobin over 28 days | Up to 28 days
  Haemoglobin concentration will be measured on peripheral blood samples (HemoCue) at baseline (before drug administration) and on Days 3, 6, 8, 15, 20 and 28.
Safety: Change in haemotocrit over 28 days | Up to 28 days
  Haematocrit will be measured at baseline (before drug administration), and on Days 3, 6, 8, 15, 20 and 28 using venous blood, that is drawn into a centrifuge tube and centrifuged to separate cellular components.
Safety: Change in methaemoglobin over 28 days | Up to 28 days
  Methaemoglobin concentration will be measured by pulse oximetry (Masimo Rad-57 Pulse CO-Oximeter with SpMet functionality) at baseline (before drug administration), and on Days 1, 3, 6, 8, 15, 20 and 28.
Safety: Change in maternal and infant weight in kilograms over 28 days | Up to 28 days
  Maternal and infant weight will be measured at all follow-up time-points (Baseline (Day 0), Days 1, 3, 6, 8, 15, 20, 28), using appropriate calibrated scales. All measurements will be recorded to the closest kilogram.
Safety: Frequency of self-reported adverse events | Up to 7 days after completion of treatment regimen
Safety: Breastfeeding behaviour | Up to 14 days
  At each follow-up time-point, mothers will be asked to report the estimated duration of breast feeding (minutes) during the previous 24 hours.
Change in alanine transaminase (ALT) over 28 days | Up to 28 days
  Alanine transaminase (ALT) will be evaluated using point-of-care biochemistry analysis (Fuji Dri-Chem NX600). Samples will be evaluated at baseline (before drug administration), and on Days 3, 6, 8, 15, 20 and 28.
Change in total bilirubin (TBil) over 28 days | Up to 28 days
  Total bilirubin (TBil) will be evaluated using point-of-care biochemistry analysis (Fuji Dri-Chem NX600). Samples will be evaluated at baseline (before drug administration) and on Days 3, 6, 8, 15, 20 and 28.
Change in creatinine (Cr) over 28 days | Up to 28 days
  Creatinine (Cr) will be evaluated using point-of-care biochemistry analysis (Fuji Dri-Chem NX600). Samples will be evaluated at at baseline (before drug administration) and on Days 3, 6, 8, 15, 20 and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Brioni Moore, PhD, Principal Investigator — Curtin University
Locations (1):
- Alexishafen Health Centre, Madang, Madang Province, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared upon contact with the principle investigators and approval by the PNG Institute of Medical Research.